CLINICAL TRIAL: NCT02979912
Title: The Use of Autologous Platelet Lysate in Persistent Corneal Epithelial Defects
Brief Title: Autologous Platelet Lysate in Corneal Epithelial Defects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hanan Jafar (Other)
Responsible Party: Sponsor-Investigator, Hanan Jafar, Researcher, University of Jordan
Organization: University of Jordan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEDUJCTC
Record Dates: First submitted 2016-11-29; First posted 2016-12-02 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Persistent Corneal Epithelial Defect
Keywords: Persistent corneal epithelial defect; Platelet Lysate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Platelet Lysate (Experimental): Autologous platelet lysate dispensed into eye droppers to be applied four times a day for a total of four weeks.
  Interventions: Biological: Platelet Lysate

INTERVENTIONS:
Biological: Platelet Lysate — Eye drops of Platelet Lysate

SUMMARY:
Patients diagnosed with persistent corneal epithelial ulcers will be treated with autologous platelet lysate.

DETAILED DESCRIPTION:
Autologous platelet lysate (PL) will be given to patients diagnosed with persistent corneal epithelial ulcers (PED) who are unresponsive to conventional therapy to promote the healing of PED. PL will be dispensed into sterile eye droppers, and these eye droppers will be stored ideally at -20C and thaw once for use, then will be kept in the refrigerator at +4C, to be taken in multiple doses.

ELIGIBILITY:
Inclusion Criteria:

1. Cognitive ability to understand and sign the consent form.
2. Corneal ulcers that did not re-epithelialise after 1 week of conventional treatment (therapeutic contact lenses, topical artificial tears, eye packs and antibiotic eye-drops).
3. Clinical indications: corneal ulcer due to caustic substances, corneal epitheliopathy, corneal lesions following cataract surgery, recurrent ulcerative keratitis, corneal lesions due to a foreign body.
4. Good compliance with the study regimen and availability for the duration of the entire study period.

Exclusion Criteria:

1. Corneal ulcers which developed tissue scars.
2. Pregnant or lactating women.

Ages: 21 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) as a result of the eye drops | 2 months
  Evaluation of the safety and tolerability of PL in the treatment of PED by monitoring any adverse event resulting from the eye drops.

SECONDARY OUTCOMES:
Assessment of the efficacy by clinical judgment | 6 months
  Efficacy of the given eye drops will be clinically evaluated by measuring the degree of healing of the epithelial defect

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah Awidi, MD, Study Director — Cell Therapy Center
Locations (1):
- Cell Therapy Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Abu-Ameerh MA, Jafar HD, Hasan MH, Al Bdour MD, Msallam M, Ababneh OH, Alhattab DM, Al-Kurdi B, Awidi AA, Awidi AS. Platelet lysate promotes re-epithelialization of persistent epithelial defects: a pilot study. Int Ophthalmol. 2019 Jul;39(7):1483-1490. doi: 10.1007/s10792-018-0968-1. Epub 2018 Jul 5. PMID 29978342